CLINICAL TRIAL: NCT02758951
Title: Perioperative Systemic Therapy and Cytoreductive Surgery with HIPEC Versus Upfront Cytoreductive Surgery with HIPEC Alone for Isolated Resectable Colorectal Peritoneal Metastases: a Multicentre, Open-label, Parallel-group, Phase II-III, Randomised Superiority Study
Brief Title: Perioperative Systemic Therapy for Isolated Resectable Colorectal Peritoneal Metastases
Acronym: CAIRO6
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Koen Rovers (Other)
Collaborators: Dutch Cancer Society (Other); Comprehensive Cancer Centre The Netherlands (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor-Investigator, Koen Rovers, Coordinating Investigator, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL57644.100.16; 2016-001865-99 (EudraCT Number); ISRCTN15977568 (Registry Identifier: ISRCTN); NTR6301 (Registry Identifier: NTR)
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Neoplasm; Colorectal Cancer; Colorectal Neoplasms Malignant; Colorectal Carcinoma; Colorectal Adenocarcinoma; Peritoneal Neoplasms; Peritoneal Carcinomatosis; Peritoneal Cancer; Peritoneal Metastases; Peritoneal Neoplasm Malignant Secondary Carcinomatosis; Peritoneal Neoplasm Malignant Secondary
Keywords: Colorectal Neoplasms; Peritoneal Neoplasms; Cytoreduction Surgical Procedures; Hyperthermia, Induced; Neoadjuvant Therapy; Adjuvant Chemotherapy; Bevacizumab; Randomized Controlled Trial; Mortality; Progression-Free Survival
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Peritoneal Neoplasms; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perioperative systemic therapy and CRS-HIPEC (Experimental): At the discretion of the treating physician, perioperative systemic therapy consists of either four 3-weekly neoadjuvant and adjuvant cycles of capecitabine with oxaliplatin (CAPOX), six 2-weekly neoadjuvant and adjuvant cycles of 5-fluorouracil/leucovorin with oxaliplatin (FOLFOX), or six 2-weekly neoadjuvant cycles of 5-fluorouracil/leucovorin with irinotecan (FOLFIRI) followed by either four 3-weekly (capecitabine) or six 2-weekly (5-fluorouracil/leucovorin) adjuvant cycles of fluoropyrimidine monotherapy. Bevacizumab is added to the first three (CAPOX) or four (FOLFOX/FOLFIRI) neoadjuvant cycles.
  CRS-HIPEC is performed according to the Dutch protocol in all study centres.
  Interventions: Other: Perioperative systemic therapy; Combination Product: Perioperative CAPOX-bevacizumab; Combination Product: Perioperative FOLFOX-bevacizumab; Combination Product: Perioperative FOLFIRI-bevacizumab; Procedure: CRS-HIPEC, experimental arm
- Upfront CRS-HIPEC alone (Active Comparator): CRS-HIPEC is performed according to the Dutch protocol in all study centres.
  Interventions: Procedure: CRS-HIPEC, control arm

INTERVENTIONS:
Other: Perioperative systemic therapy — Neoadjuvant systemic therapy should start within four weeks after randomisation. Adjuvant systemic therapy should start within twelve weeks after CRS-HIPEC. In case of unacceptable toxicity or contraindications to oxaliplatin or irinotecan in the neoadjuvant setting, CAPOX or FOLFOX may be switched to FOLFIRI and vice versa. In case of unacceptable toxicity or contraindications to oxaliplatin in the adjuvant setting, CAPOX of FOLFOX may be switched to fluoropyrimidine monotherapy. Dose reduction, prohibited concomitant care, permitted concomitant care, and strategies to improve adherence are not specified a priori, but left to the discretion of the treating medical oncologist. Perioperative systemic therapy can be prematurely discontinued due to radiological or clinical disease progression, unacceptable toxicity, physicians decision, or at patients request.
  Arms: Perioperative systemic therapy and CRS-HIPEC
Combination Product: Perioperative CAPOX-bevacizumab — Four three-weekly neoadjuvant and adjuvant cycles of CAPOX (130 mg/m2 body-surface area [BSA] of oxaliplatin, intravenously [IV] on day 1; 1000 mg/m2 BSA of capecitabine, orally twice daily on days 1-14), with bevacizumab (7.5 mg/kg body weight, IV on day 1) added to the first three neoadjuvant cycles.
  Arms: Perioperative systemic therapy and CRS-HIPEC
Combination Product: Perioperative FOLFOX-bevacizumab — Six two-weekly neoadjuvant and adjuvant cycles of FOLFOX (85 mg/m2 body-surface area [BSA] of oxaliplatin, intravenously [IV] on day 1; 400 mg/m2 BSA of leucovorin, IV on day 1; 400/2400 mg/m2 BSA of bolus/continuous 5-fluorouracil, IV on day 1-2), with bevacizumab (5 mg/kg body weight, IV on day 1) added to the first four neoadjuvant cycles.
  Arms: Perioperative systemic therapy and CRS-HIPEC
Combination Product: Perioperative FOLFIRI-bevacizumab — Six two-weekly neoadjuvant cycles of FOLFIRI (180 mg/m2 body-surface area [BSA] of irinotecan, intravenously [IV] on day 1; 400 mg/m2 BSA of leucovorin, IV on day 1; 400/2400 mg/m2 BSA of bolus/continuous 5-fluorouracil, IV on day 1-2) and either four three-weekly (capecitabine (1000 mg/m2 BSA, orally twice daily on days 1-14) or six two-weekly (400 mg/m2 BSA of leucovorin, IV on day 1; 400/2400 mg/m2 BSA of bolus/continuous 5-fluorouracil, IV on day 1-2) adjuvant cycles of fluoropyrimidine monotherapy, with bevacizumab (5 mg/kg body weight, IV on day 1) added to the first four neoadjuvant cycles.
  Arms: Perioperative systemic therapy and CRS-HIPEC
Procedure: CRS-HIPEC, experimental arm — CRS-HIPEC is performed according to the Dutch protocol in all study centres. Until publication of the PRODIGE7 trial, the choice of HIPEC medication (oxaliplatin or mitomycin C) has been left to the discretion of the treating physician, since neither one had a favourable safety or efficacy until then. After publication of the PRODIGE7 trial in 2021, oxaliplatin-based HIPEC was omitted in all centres (and therefore automatically omitted in the present study), and all centres switched to mitomycin C-based HIPEC. CRS-HIPEC should be performed within six weeks after completion of neoadjuvant systemic therapy in case of sufficient clinical condition, and at least six weeks after the last administration of bevacizumab in order to minimise the risk of bevacizumab-related postoperative complications.
  Arms: Perioperative systemic therapy and CRS-HIPEC
Procedure: CRS-HIPEC, control arm — CRS-HIPEC is performed according to the Dutch protocol in all study centres. Until publication of the PRODIGE7 trial, the choice of HIPEC medication (oxaliplatin or mitomycin C) has been left to the discretion of the treating physician, since neither one had a favourable safety or efficacy until then. After publication of the PRODIGE7 trial in 2021, oxaliplatin-based HIPEC was omitted in all centres (and therefore automatically omitted in the present study), and all centres switched to mitomycin C-based HIPEC. CRS-HIPEC should be performed within six weeks after randomisation.
  Arms: Upfront CRS-HIPEC alone

SUMMARY:
This is a multicentre, open-label, parallel-group, phase II-III, superiority study that randomises patients with isolated resectable colorectal peritoneal metastases in a 1:1 ratio to receive either perioperative systemic therapy and cytoreductive surgery with HIPEC (experimental arm) or upfront cytoreductive surgery with HIPEC alone (control arm).

DETAILED DESCRIPTION:
Rationale: cytoreductive surgery with HIPEC (CRS-HIPEC) is a curative intent treatment for patients with isolated resectable colorectal peritoneal metastases (PM). Upfront CRS-HIPEC alone is the standard treatment in the Netherlands. The addition of neoadjuvant and adjuvant systemic therapy (together: perioperative systemic therapy) to CRS-HIPEC could have benefits and drawbacks. Potential benefits are eradication of systemic micrometastases, preoperative intraperitoneal tumour downstaging, elimination of post-surgical residual cancer cells, and improved patient selection for CRS-HIPEC. Potential drawbacks are preoperative disease progression and secondary unresectability for CRS-HIPEC, systemic therapy related toxicity, increased postoperative morbidity, decreased quality of life, and higher costs. Currently, there is a complete lack of randomised studies that prospectively compare the oncological efficacy of perioperative systemic therapy and CRS-HIPEC with upfront CRS-HIPEC alone. Notwithstanding this lack of evidence, perioperative systemic therapy is widely administered to patients with isolated resectable colorectal PM. However, administration and timing of perioperative systemic therapy vary substantially between countries, hospitals, and guidelines. More importantly, it remains unknown whether perioperative systemic therapy has an intention-to-treat benefit in this setting. Therefore, this study randomises patients with isolated resectable colorectal PM to receive either perioperative systemic therapy (experimental arm) or upfront CRS-HIPEC alone (control arm).

Study design: a multicentre, open-label, parallel-group, phase II-III, superiority study that randomises eligible patients in a 1:1 ratio.

Objectives: objectives of the phase II study (80 patients) are to explore the feasibility of accrual, the feasibility, safety, and tolerance of perioperative systemic therapy, and the radiological and pathological response of colorectal PM to neoadjuvant systemic therapy. The primary objective of the phase III study (358 patients) is to compare overall survival between both arms. Secondary objectives are to assess progression-free and disease-free survival, surgical characteristics, major postoperative morbidity, patient-reported outcomes, and costs in both arms. Other objectives are to assess major systemic therapy related toxicity and the objective radiological and pathological response of colorectal PM to neoadjuvant systemic therapy.

Study population: adults who have a good performance status, histological or cytological proof of PM of a colorectal adenocarcinoma, resectable disease, no systemic colorectal metastases within three months prior to enrolment, no systemic therapy for colorectal cancer within six months prior to enrolment, no previous CRS-HIPEC, no contraindications for the planned systemic treatment or CRS-HIPEC, and no relevant concurrent malignancies.

Intervention: at the discretion of the treating medical oncologist, perioperative systemic therapy consists of either four 3-weekly neoadjuvant and adjuvant cycles of capecitabine with oxaliplatin (CAPOX), six 2-weekly neoadjuvant and adjuvant cycles of 5-fluorouracil/leucovorin with oxaliplatin (FOLFOX), or six 2-weekly neoadjuvant cycles of 5-fluorouracil/leucovorin with irinotecan (FOLFIRI) followed by either four 3-weekly (capecitabine) or six 2-weekly (5-fluorouracil/leucovorin) adjuvant cycles of fluoropyrimidine monotherapy. Bevacizumab is added to the first three (CAPOX) or four (FOLFOX/FOLFIRI) neoadjuvant cycles.

Endpoints: primary endpoints of the phase II study are to explore the feasibility and safety of perioperative systemic therapy by comparing proportions of patients undergoing complete CRS-HIPEC and proportions of patients with major postoperative morbidity between both arms. The primary comparative endpoint of the phase III study is overall survival. Major secondary endpoints assessed in both arms are proportions of major postoperative morbidity, progression-free survival, disease-free survival, patient-reported outcomes (PROs), and costs. Major secondary endpoints assessed in the experimental arm are the proportion of patients with major systemic therapy related toxicity and the proportions of patients with objective radiological and pathological responses of colorectal PM to neoadjuvant systemic therapy.

Statistical analysis: the study is powered to detect an increase in 3-year overall survival from 50% in the control arm to 65% in the experimental arm (corresponding hazard ratio 0.62), which is considered to be a clinically relevant difference by the investigators. A total number of 358 patients (179 in each arm) is needed to detect this hypothesized difference with 5% drop-out, 80% power, and a two-sided log-rank test of p<0.05. In August 2024, when several patients in the experimental arm were still receiving trial treatment, a regular follow-up update revealed that 156 events for the primary outcome (i.e. deaths) had occurred. The study then had 85% power to detect the hypothesized hazard ratio of 0.62 for overall survival in the analysis of superiority of the experimental arm relative to the control arm at a two-sided alpha of 0.05. After discussing these data with the Data Monitoring Committee and the medical ethics committee, it was decided to schedule data cut-off for a first analysis of the primary outcome at the time the last patient in the experimental arm (enrolled April 2024) finishes trial treatment, which is expected 1 November 2024 at an estimated number of +/- 172 events (+/- 88% power).

ELIGIBILITY:
Eligible patients are adults who have:

* a World Health Organisation (WHO) performance status of ≤1;
* histological or cytological proof of PM of a non-appendiceal colorectal adenocarcinoma with ≤50% of the tumour cells being signet ring cells;
* resectable disease determined by a diagnostic laparoscopy/laparotomy in combination with abdominal computed tomography and/or magnetic resonance imaging (MRI); only in patients in whom diagnostic laparoscopy or laparotomy is considered not feasible or valuable (e.g. due to known adhesions impeding adequate PCI scoring), it is also allowed to determine resectability by CT or MRI only (provided that the colorectal PM are histologically or cytologically proven);
* no evidence of systemic colorectal metastases within three months prior to enrolment;
* no systemic therapy for colorectal cancer within six months prior to enrolment;
* no contraindications for CRS-HIPEC;
* no previous CRS-HIPEC;
* no concurrent malignancies that interfere with the planned study treatment or the prognosis of resected colorectal PM.

Importantly, enrolment is allowed for patients with radiologically non-measurable disease. Enrolment is also allowed for patients who are referred to a study centre after a macroscopically complete resection of colorectal PM in a referring centre, since it is assumed that microscopic (and often macroscopic) colorectal PM are still present. The diagnostic laparoscopy/laparotomy may be performed in a referring centre, provided that the peritoneal cancer index (PCI) is appropriately scored and documented before enrolment.

Patients are excluded in case of any comorbidity or condition that prevents safe administration of the planned perioperative systemic therapy, determined by the treating medical oncologist, e.g.:

* Inadequate bone marrow, renal, or liver functions (e.g. haemoglobin <6.0 mmol/L, neutrophils <1.5 x 109/L, platelets <100 x 109/L, serum creatinine >1.5 x ULN, creatinine clearance <30 ml/min, bilirubin >2 x ULN, serum liver transaminases >5 x ULN);
* Previous intolerance of fluoropyrimidines or both oxaliplatin and irinotecan;
* Dehydropyrimidine dehydrogenase deficiency;
* Serious active infections;
* Severe diarrhoea;
* Stomatitis or ulceration in the mouth or gastrointestinal tract;
* Recent major cardiovascular events;
* Unstable or uncompensated respiratory or cardiac disease;
* Bleeding diathesis or coagulopathy;
* Pregnancy or lactation.

The aforementioned laboratory values and tests are to be determined at the discretion of the physician, e.g. only if the patient is suspect for abnormal conditions tests will be conducted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From enrolment up to five years thereafter
  Time between enrolment and death due to any cause

SECONDARY OUTCOMES:
Progression-free survival | From enrolment up to five years thereafter
  Time between enrolment and physician-determined disease progression before CRS-HIPEC, CRS-HIPEC in case of unresectable disease or incomplete CRS, physician-determined recurrence after CRS-HIPEC, or death due to any cause;
Disease-free survival | From enrolment up to five years thereafter
  Time between macroscopic complete CRS-HIPEC and physician-determined recurrence or death due to any cause
Macroscopic complete CRS-HIPEC | From enrolment up to approximately six weeks (control arm) or five months (experimental arm) thereafter
  The proportion of patients undergoing macroscopic complete CRS-HIPEC
Surgical characteristics: peritoneal cancer index | During CRS-HIPEC, one to five months after enrolment
  The peritoneal cancer index during explorative laparotomy
Surgical characteristics: bowel anastomoses | During CRS-HIPEC, , one to five months after enrolment
  The proportion of patients with a bowel anastomosis during CRS-HIPEC
Surgical characteristics: ostomy formations | During CRS-HIPEC, one to five months after enrolment
  The proportion of patients with an ostomy formation during CRS-HIPEC
Surgical characteristics: operating time | During CRS-HIPEC, one to five months after enrolment
  The operating time of CRS-HIPEC
Major postoperative morbidity | From (intended) CRS-HIPEC up to three months postoperatively
  The proportions of patients with Clavien-Dindo grade 3 or higher, grade 4 or higher, and grade 5 postoperative morbidity
Postoperative hospital stay | During the postoperative course of CRS-HIPEC, up to 90 days postoperatively
  The number of days between (intended) CRS-HIPEC and initial discharge
Postoperative readmissions | From CRS-HIPEC to 90 days postoperatively
  The proportion of patients with a readmission within 90 days after (intended) CRS-HIPEC
Patient-reported outcomes: EQ-5D-5L | From enrolment up to five years thereafter
  Extracted from EQ-5D-5L questionnaire at different points in time
Patient-reported outcomes: QLQ-C30 | From enrolment up to five years thereafter
  Extracted from EORTC QLQ-C30 questionnaires at different points in time
Patient-reported outcomes: QLQ-CR29 | From enrolment up to five years thereafter
  Extracted from EORTC QLQ-CR29 questionnaire at different points in time
Costs | From enrolment up to five years thereafter
  Extracted from questionnaire (iMTA PCQ, iMTA MCQ) at different points in time

OTHER OUTCOMES:
Major systemic therapy-related toxicity (experimental arm) | From the first administration of systemic therapy up to 30 days after the last administration
  Proportions of patients with CTCAE grade 3 or higher, grade 4 or higher, and grade 5 systemic therapy-related toxicity
Radiological response to neoadjuvante treatment (experimental arm) | After radiological restaging during neoadjuvant treatment, approximately three months after randomisation
  The proportion of patients with an objective radiological response of colorectal peritoneal metastases to neoadjuvant systemic therapy, determined by central review of thoracoabdominal CTs before and after neoadjuvant treatment by two radiologists blinded for clinical outcomes. Radiological response is assessed according to (1) standard RECIST criteria and (2) the radiological PCI. Response according to radiological PCI is classified as complete response (i.e. disappearance of all peritoneal lesions), partial response (i.e. ≥30% decrease of PCI), stable disease (i.e. <30% decrease or <20% increase of PCI), progressive disease (i.e. ≥20% increase of PCI), or non-evaluable. When in situ, the primary tumour is not included in response assessment according to the radiological PCI.
Pathological response to neoadjuvant treatment (experimental arm) | After (intended) CRS-HIPEC, approximately five months after randomisation
  The proportion of patients with an objective pathological response of colorectal peritoneal metastases to neoadjuvant systemic therapy, determined by central review of resected specimens during CRS-HIPEC by two pathologists blinded for clinical outcomes. Pathological response is assessed using (1) the peritoneal regression grading score (PRGS) and (2) the standard Mandard tumour regression grading (TRG).

CONTACTS AND LOCATIONS:
Overall Officials: Ignace H de Hingh, MD, PhD, Study Chair — Catharina Hospital, Eindhoven, Netherlands; Pieter J Tanis, MD, PhD, Study Director — Department of Surgery, Amsterdam University Medical Centre, Location AMC, Amsterdam, Netherlands; Cornelis J Punt, MD, PhD, Study Director — Department of Medical Oncology, Amsterdam University Medical Centre, Location AMC, Amsterdam, Netherlands; Alexandra R Brandt-Kerkhof, MD, Principal Investigator — Department of Surgery, Erasmuc University Medical Centre, Rotterdam, Netherlands; Jurriaan B Tuynman, MD, PhD, Principal Investigator — Department of Surgery, Amsterdam University Medical Centre, Location VUMC, Amsterdam, Netherlands; Arend G Aalbers, MD, Principal Investigator — Department of Surgery, Netherlands Cancer Institute, Amsterdam, Netherlands; Marinus J Wiezer, MD, PhD, Principal Investigator — Department of Surgery, St. Antonius Hospital, Nieuwegein, Netherlands; Patrick H Hemmer, MD, Principal Investigator — Department of Surgery, University Medical Centre Groningen, Groningen, Netherlands; Sandra A Radema, MD, PhD, Principal Investigator — Department of Medical Oncology, Radboud University Medical Centre, Nijmegen, Netherlands; Wilhemina M van Grevenstein, MD, PhD, Principal Investigator — Department of Surgery, University Medical Centre Utrecht, Utrecht, Netherlands; Eino B van Duyn, MD, PhD, Principal Investigator — Department of Surgery, Medisch Spectrum Twente, Enschede, Netherlands; Ignace H de Hingh, MD, PhD, Principal Investigator — Department of Surgery, Catharina Hospital, Eindhoven, Netherlands
Locations (9):
- Ziekenhuis Oost-Limburg, Genk, Flanders, Belgium
- Netherlands (8):
  - Amsterdam University Medical Centre, Location VUMC, Amsterdam
  - Netherlands Cancer Institute, Amsterdam
  - Catharina Hospital, Eindhoven
  - University Medical Centre Groningen, Groningen
  - St. Antonius Hospital, Nieuwegein
  - Radboud University Medical Centre, Nijmegen
  - Erasmus University Medical Centre, Rotterdam
  - University Medical Centre Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
The full protocol and Dutch informed consent forms are publicly accessible (https://dccg.nl/trial/cairo-6). Participant-level datasets and statistical codes will become available upon reasonable request after the results of the study have been published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The full protocol and Dutch informed consent forms are publicly accessible (https://dccg.nl/trial/cairo-6). Participant-level datasets and statistical codes will become available upon reasonable request after the results of the study have been published.
Access Criteria: Reasonable request.

REFERENCES:
- [Background] Rovers KP, Bakkers C, Nienhuijs SW, Burger JWA, Creemers GM, Thijs AMJ, Brandt-Kerkhof ARM, Madsen EVE, van Meerten E, Tuynman JB, Kusters M, Versteeg KS, Aalbers AGJ, Kok NFM, Buffart TE, Wiezer MJ, Boerma D, Los M, de Reuver PR, Bremers AJA, Verheul HMW, Kruijff S, de Groot DJA, Witkamp AJ, van Grevenstein WMU, Koopman M, Nederend J, Lahaye MJ, Kranenburg O, Fijneman RJA, van 't Erve I, Snaebjornsson P, Hemmer PHJ, Dijkgraaf MGW, Punt CJA, Tanis PJ, de Hingh IHJT; Dutch Peritoneal Oncology Group and the Dutch Colorectal Cancer Group. Perioperative Systemic Therapy vs Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy Alone for Resectable Colorectal Peritoneal Metastases: A Phase 2 Randomized Clinical Trial. JAMA Surg. 2021 Aug 1;156(8):710-720. doi: 10.1001/jamasurg.2021.1642. PMID 34009291
- [Background] Rovers KP, Bakkers C, Simkens GAAM, Burger JWA, Nienhuijs SW, Creemers GM, Thijs AMJ, Brandt-Kerkhof ARM, Madsen EVE, Ayez N, de Boer NL, van Meerten E, Tuynman JB, Kusters M, Sluiter NR, Verheul HMW, van der Vliet HJ, Wiezer MJ, Boerma D, Wassenaar ECE, Los M, Hunting CB, Aalbers AGJ, Kok NFM, Kuhlmann KFD, Boot H, Chalabi M, Kruijff S, Been LB, van Ginkel RJ, de Groot DJA, Fehrmann RSN, de Wilt JHW, Bremers AJA, de Reuver PR, Radema SA, Herbschleb KH, van Grevenstein WMU, Witkamp AJ, Koopman M, Haj Mohammad N, van Duyn EB, Mastboom WJB, Mekenkamp LJM, Nederend J, Lahaye MJ, Snaebjornsson P, Verhoef C, van Laarhoven HWM, Zwinderman AH, Bouma JM, Kranenburg O, van 't Erve I, Fijneman RJA, Dijkgraaf MGW, Hemmer PHJ, Punt CJA, Tanis PJ, de Hingh IHJT; Dutch Peritoneal Oncology Group (DPOG); Dutch Colorectal Cancer Group (DCCG). Perioperative systemic therapy and cytoreductive surgery with HIPEC versus upfront cytoreductive surgery with HIPEC alone for isolated resectable colorectal peritoneal metastases: protocol of a multicentre, open-label, parallel-group, phase II-III, randomised, superiority study (CAIRO6). BMC Cancer. 2019 Apr 25;19(1):390. doi: 10.1186/s12885-019-5545-0. PMID 31023318
- [Derived] Peng S, Chen D, Cai J, Yuan Z, Huang B, Li Y, Wang H, Luo Q, Kuang Y, Liang W, Liu Z, Wang Q, Cui Y, Wang H, Liu X. Enhancing cancer-associated fibroblast fatty acid catabolism within a metabolically challenging tumor microenvironment drives colon cancer peritoneal metastasis. Mol Oncol. 2021 May;15(5):1391-1411. doi: 10.1002/1878-0261.12917. Epub 2021 Feb 16. PMID 33528867
- See also: Related Info — https://dccg.nl/trial/cairo-6